CLINICAL TRIAL: NCT01619826
Title: Enhancing Children's Cognitive and Brain Health Through Physical Activity Training
Brief Title: Enhancing Children's Cognitive and Brain Health Through Physical Activity Training (FITKids2)
Acronym: FITKids2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HD069381; R01HD069381-01A1 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cognitive Ability, General; Achievement
Keywords: physical activity; fitness; brain health; cognition; scholastic achievement; preadolescent children
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Participants randomized to the physical activity-based afterschool intervention
  Interventions: Behavioral: Physical Activity
- Wait List Group (Placebo Comparator): Participants in this group partake in their regular afterschool activities, without intervention from the study staff.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 9-month afterschool program designed to increase physical activity and aerobic fitness.
  Arms: Treatment Group
Behavioral: Physical Activity — Participants in this group partake in their regular afterschool activities, without intervention from the study staff.
  Arms: Wait List Group

SUMMARY:
The objective of this study is to use a randomized controlled design to determine whether cardiorespiratory fitness training improves neurocognitive function and academic performance during preadolescent development.

DETAILED DESCRIPTION:
The long term objective of this project is to develop an understanding of lifestyle factors that influence the cognitive and brain health of children while also reducing the sedentary nature of today's youth. Previous research has found that physical activity interventions can enhance both a variety of aspects of cognition and brain structure and function of children, older adults, and individuals with neurodegenerative disorders such as Parkinson's disease and multiple sclerosis. More specifically, in previous research with children the researchers have found that higher fit children possess larger hippocampi which in turn are related to better relational memory than their lower fit counterparts. The researchers have also observed that higher fit children exhibit more efficient executive control as indicated by performance measures and event-related brain potentials. While intriguing, these cross-sectional data do not enable us to establish causality between physical activity and cognition. In the current study the researchers substantially extend this previous research by examining the influence of a 9 month randomized controlled afterschool physical activity program on cognition and brain health. Cognition will be assessed with a battery of tasks and standardized achievement tests both before and after the 9 month intervention in the activity group and a wait list control (who will receive the intervention the following year). Children will also participate in magnetic resonance imaging (MRI) sessions both before and after the intervention (and at comparable times for the wait list control). In these sessions the researchers will measure both structural aspects of the brain including regional volumes of gray matter and the integrity of the white matter tracts (through diffusion tensor imaging) and functional aspects of brain function using fMRI activity recorded as the children perform a series of executive control and memory tasks. The researchers anticipate, based on our cross-sectional studies with children and our previous longitudinal studies with older adults, that the children in the physical activity program will show both larger regional brain volumes, particularly in brain regions that subserve executive control and relational memory, and more efficient brain function, as indexed by task-related and resting state fMRI. Furthermore, the researchers anticipate that these changes will be accompanied by improvements in memory and executive control processes. Given recent trends identifying decreased levels of physical activity and health status in preadolescents, the understanding of the potential benefits of physical activity on cognition is of great interest. It is imperative that factors positively influencing cognitive function of children be examined to maximize health and effective functioning of individuals as they progress through the lifespan.

ELIGIBILITY:
Inclusion Criteria:

* Parental/guardian consent
* 8 - 9 years old
* Capable of performing exercise
* Absence of school-identified learning disability
* IQ >= 85
* Tanner Scales score <= 2
* ADHD Rating Scales score >= 85%
* Right hand dominant
* Absence of metal implants
* Not claustrophobic

Exclusion Criteria:

* Non-consent of guardian
* Above or below 8 - 9 years old
* Any physical disability that prohibits exercise
* School-identified learning disability
* IQ < 85
* Tanner Scales score > 2
* ADHD Rating Scale score < 85%
* Left hand dominant
* Presence of metal implants
* Claustrophobic

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
NeuroCognitive Assessment | Change from baseline, 36 - 40 weeks
  Normed computerized test battery for cognitive testing
Structural Magnetic Resonance Imaging | Change from baseline, 36 - 40 weeks
  Measures of brain structure
Functional Magnetic Resonance Imaging | Change from baseline, 36 - 40 weeks
  Measures of brain function
Academic Achievement | Change from baseline, 36 - 40 weeks
  Scholastic achievement tests of reading comprehension and arithmetic
Eye Tracking | Change from baseline, 36 - 40 weeks
  Measures of visual gaze
Task Performance | Change from baseline, 36 - 40 weeks
  Measures of responses speed and accuracy

SECONDARY OUTCOMES:
Event-related Brain Potentials | Change from baseline, 36 - 40 weeks
  Measures of the neuroelectric system that occur in response to, or in preparation for, a discrete event
DXA Body Mass Assessment | Change from baseline, 36 - 40 weeks
  Measures of bone density, total body composition, and fat content
Diet and Brain Function | Change from baseline, 36-40 weeks
  Measure of correlation between diet and brain function
Adiposity | Change from baseline, 36 - 40 weeks
  Measure of change in adiposity

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Kramer, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Charles Hillman, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (4):
- United States (4):
  - Beckman Institute - Biomedical Imaging Center, Urbana, Illinois
  - Campus Recreation Center East, Urbana, Illinois
  - Department of Kinesiology and Community Health, Urbana, Illinois
  - University of Illinois at Urbana-Champaign, Urbana, Illinois

REFERENCES:
- [Derived] Liu R, Hannon BA, Robinson KN, Raine LB, Hammond BR, Renzi-Hammond LM, Cohen NJ, Kramer AF, Hillman CH, Teran-Garcia M, Khan NA. Single Nucleotide Polymorphisms in CD36 Are Associated with Macular Pigment among Children. J Nutr. 2021 Sep 4;151(9):2533-2540. doi: 10.1093/jn/nxab153. PMID 34049394
- [Derived] Chojnacki MR, Holscher HD, Balbinot AR, Raine LB, Biggan JR, Walk AM, Kramer AF, Cohen NJ, Hillman CH, Khan NA. Relations between mode of birth delivery and timing of developmental milestones and adiposity in preadolescence: A retrospective study. Early Hum Dev. 2019 Feb;129:52-59. doi: 10.1016/j.earlhumdev.2018.12.021. Epub 2019 Jan 12. PMID 30641478
- [Derived] Chojnacki MR, Raine LB, Drollette ES, Scudder MR, Kramer AF, Hillman CH, Khan NA. The Negative Influence of Adiposity Extends to Intraindividual Variability in Cognitive Control Among Preadolescent Children. Obesity (Silver Spring). 2018 Feb;26(2):405-411. doi: 10.1002/oby.22053. Epub 2017 Dec 27. PMID 29282881
- [Derived] Raine LB, Khan NA, Drollette ES, Pontifex MB, Kramer AF, Hillman CH. Obesity, Visceral Adipose Tissue, and Cognitive Function in Childhood. J Pediatr. 2017 Aug;187:134-140.e3. doi: 10.1016/j.jpeds.2017.05.023. Epub 2017 Jun 13. PMID 28622956
- [Derived] Barnett SM, Khan NA, Walk AM, Raine LB, Moulton C, Cohen NJ, Kramer AF, Hammond BR Jr, Renzi-Hammond L, Hillman CH. Macular pigment optical density is positively associated with academic performance among preadolescent children. Nutr Neurosci. 2018 Nov;21(9):632-640. doi: 10.1080/1028415X.2017.1329976. Epub 2017 May 23. PMID 28535707
- [Derived] Hassevoort KM, Khazoum SE, Walker JA, Barnett SM, Raine LB, Hammond BR, Renzi-Hammond LM, Kramer AF, Khan NA, Hillman CH, Cohen NJ. Macular Carotenoids, Aerobic Fitness, and Central Adiposity Are Associated Differentially with Hippocampal-Dependent Relational Memory in Preadolescent Children. J Pediatr. 2017 Apr;183:108-114.e1. doi: 10.1016/j.jpeds.2017.01.016. Epub 2017 Feb 8. PMID 28189300
- [Derived] Baym CL, Khan NA, Monti JM, Raine LB, Drollette ES, Moore RD, Scudder MR, Kramer AF, Hillman CH, Cohen NJ. Dietary lipids are differentially associated with hippocampal-dependent relational memory in prepubescent children. Am J Clin Nutr. 2014 May;99(5):1026-32. doi: 10.3945/ajcn.113.079624. Epub 2014 Feb 12. PMID 24522447
- See also: FITKids Website — http://labs.kch.illinois.edu/Research/Labs/neurocognitive-kinesiology/outreach/fitkids/default.htm